CLINICAL TRIAL: NCT00776802
Title: Phase 1/2 Study of GCS-100 in Combination With Etoposide and Dexamethasone in Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: GCS-100LE in Combination With Etoposide and Dexamethasone in Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: GCS-100LE
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-CS010
Record Dates: First submitted 2008-10-19; First posted 2008-10-21 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: GCS-100; Diffuse Large B-cell Lymphoma; DLBCL; Relapsed or refractory DLBCL; Etoposide; Dexamethasone
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — GCS-100; Etoposide; Dexamethasone; etoposide phosphate; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GCS-10 (Experimental)
  Interventions: Drug: GCS-100; Drug: Etoposide; Dexamethasone

INTERVENTIONS:
Drug: GCS-100 — GCS-100 80 mg/m2 IV (in the vein) on Study Days 1, 2, 3, 4, and 5 of a 21-day course. Three or up to six patients will be enrolled in each cohort until the maximum tolerated dose is reached. The dose levels: 1) 80 mg/m2; 2) 120 mg/m2; 3) 160 mg/m2
Drug: Etoposide; Dexamethasone — Etoposide 100 mg/m2 on Study Days 3, 4 and 5; Dexamethasone 10 mg/m2 on Study Days 1, 2, 3, 4 and 5.
  Other Names: Eposin; VP-16; Etopophos; Vepesid; Decadron

SUMMARY:
Phase 1/2, open-label, dose-escalation study to assess the safety and tolerability of GCS-100 in combination with etoposide and dexamethasone in patients with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This study will investigate the safety and efficacy of the combination of GCS-100 with etoposide and dexamethasone. In vitro data demonstrates potentiation of the killing of lymphoma cells when GCS-100 is combined with dexamethasone or etoposide (Linda Baum, unpublished data; Finbarr Cotter et al, Annals of Oncology, vol 16, 205, Suppl 5.) GCS-100 will be administered in increasing doses to define a maximum tolerated dose (MTD) in combination with these chemotherapeutic agents. When the MTD is defined, the cohort will be expanded to characterize the efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 18 years of age or older with diffuse large B-cell cell lymphoma (DLBCL) relapsed or refractory after initial therapy who:

  * Are not candidates for autologous stem cell transplant.
  * Have relapsed after autologous or allogeneic stem cell transplant.
  * Have relapsed or refractory disease after 3 successive chemotherapy regimens.
* ECOG Performance Score 0-2
* Creatinine clearance > 60 mL/min/1.73 m2.
* Total bilirubin ≤2.0 X Institutional Upper Limit of Normal (IULN)
* AST (SGOT)/ALT (SGPT) ≤2.5 X IUNL, or ≤5X IUNL in patients with liver involvement of DLBCL
* Absolute neutrophil count >1,000 /_L; hemoglobin >9 g/mL; platelet count > 75,000 /_L at screening.
* Patients must be capable of understanding the purpose and risks of the study and able to provide written consent.
* Patients must be willing and able to comply with the prescribed treatment protocol and evaluations

Exclusion Criteria:

* Treatment with experimental (unlicensed) drug within 3 weeks of treatment.
* Previous chemotherapy, or major surgery within 21 days prior to first study treatment, or radiation therapy within 6 weeks.
* Rapidly progressive disease or organ function threatened by disease
* Serious, uncontrolled active infections.
* Serologically positive for HIV, HBV, or HCV.
* Clinically significant cardiac, pulmonary, and/or hepatic dysfunction
* Lymphoma involving the central nervous system
* Female patients who are pregnant or breast feeding.
* Patients not capable of understanding the purpose and risks of the study and or unable to provide written consent.
* Patients not willing and or unable to comply with the prescribed treatment protocol and evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of GCS-100 in combination with etoposide and dexamethasone by comprehensive lab, pharmacokinetics, physical assessments, and PET-CT imaging. | Study Day 12 for toxicity, and 21-day cycles assessed every 2 cycles by physical and imaging assessments until disease progression

SECONDARY OUTCOMES:
Overall response rate; correlate response to GCS-100 with the expression of galectin-3 in tumors; correlate serum galectin-3 levels with the administration of GCS-100 | Baseline, Day 1, and Day 5 laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Pinter-Brown, MD, Principal Investigator — UCLA, Division of Hematology/Oncology
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States